CLINICAL TRIAL: NCT06008496
Title: The POPPY Study: Patient Reported Outcomes, Postoperative Pain and Pain Relief After Day Case Surgery
Brief Title: Patient Reported Outcomes, Postoperative Pain and Pain Relief After Day Case Surgery (POPPY)
Acronym: POPPY
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: National Institute for Academic Anaesthesia (Unknown); Newcastle PROMS (Unknown); Research and Audit Federation of Anaesthetic Trainees (RAFT) (Unknown); University of Plymouth (Other)
Responsible Party: Sponsor
Other Study IDs: 23/SED/793
Record Dates: First submitted 2023-05-02; First posted 2023-08-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pain; Post Operative Pain; Opioid Use; Chronic Pain
MeSH Terms: conditions — Pain; Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Day case surgery — Operation, surgical group, magnitude of surgery, anaesthetic type.

SUMMARY:
Around 3 out of 4 operations in the UK are performed as day-case, meaning the patient goes home on the same day of their operation. Hospitals usually do not follow up patients after day-case operations so we do not know very much about their short or long-term recovery. Some patients, even those who have had small operations, can develop persistent pain afterwards that continues for a long time (months to years). These patients may end up taking strong painkillers for a long time and this risks serious side effects and long-term health problems.

The POPPY study aims to find out what recovery from day-case operations is like from the patient's point of view. We will look at the first week after patients' operations and then at 3 months to see if they are in pain, and if so what pain relief they are taking.

All adults over the 5-day study period having day-case operations in the UK, with an anaesthetist, will be eligible if they have access to a smartphone. Patients will be recruited on the day of their operation from over 100 NHS hospitals. Some relevant information about the patient's current health, operation and anaesthetic will be recorded from their notes. Afterwards participants will get a text message at days 1, 3 and 7 and the at 3 months. These will connect to a data secure online questionnaire about pain, recovery, and what medications they are taking. A small number of participants with ongoing pain at 3 months will be invited to take part in a structured interview to understand their experience in more depth.

This study will provide important information that may be used to improve care of patients having day-case operations and plan future research studies aimed to prevent persistent pain and long-term use of strong painkillers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older on day of surgery
* Day-case surgery as defined by National Day Surgery Delivery Pack (NEED REF)
* An anaesthetist must be present for case.
* The procedure must involve one or more of: sedation, regional anaesthesia, central neuraxial anaesthesia or general anaesthesia

Exclusion Criteria:

* Less than 18 years of age on day of surgery
* No anaesthetist involved with the procedure (such as local anaesthesia provided by a surgeon)
* Overnight stay (admission to hospital)
* Participant lacking capacity for consent
* Diagnostic and/or minimally invasive procedures (e.g., radiology, endoscopy, or cardiology procedures)
* Pregnancy or obstetric related procedures (pregnancy per-se is not an exclusion criterion).
* Currently breast feeding
* Ophthalmic procedures
* No access to Smartphone and email
* Prisoners

Eligibility for qualitative component:

As above, plus reporting PPSP and/or PPOU at day 97 post operative

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing day-case surgery in the UK
Sampling Method: Non-Probability Sample
Enrollment: 7839 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
To measure short and long-term patient reported outcomes in UK day-case surgery patients. | 3 months
  See below outcomes for specifics (this is an overarching outcome which is broken down in the outcomes described below).
Short-term: to describe the quality of recovery over the first postoperative week | 1 week
  QOR-15 score (quality of recovery-15 score); BPI (brief pain inventory) derived pain scores; FPS (functional pain score)
Long-term: to establish the prevalence of persistent postsurgical pain (PPSP) and persistent postoperative opioid use (PPOU) in day case surgical patients. | 3 months
  PPOU prevalence (from medication use); pain at surgical site questionnaire; GAD-7 Score (generalised anxiety and depression 7 score); EQ-5D-5L score; BPI score; PHQ-8 Score (Patient Health Questionnaire 8)

SECONDARY OUTCOMES:
To identify those patient, medication, anaesthetic, and surgical characteristics that are associated with poor quality of recovery, and PPSP and/or PPOU | 3 months
  Baseline data collection: age, sex, operation type, anaesthetic type, baseline medications and medication use on day 1, 3, 7 and 97 post-op. Medication use recorded as frequency of use and medication type.
To describe the acute pain experience and analgesia use in the first postoperative week | 1 week
  BPI (brief pain inventory) score on days 1, 3, 7; analgesia medication use on days 1, 3, 7
To estimate the need for further healthcare support in the first postoperative week | 1 week
  Yes/no question on questionnaire on day 7
To determine the patient reported acceptability of SMS prompted follow-up | 1 week
  Acceptability question on questionnaire on day 7
To determine the difference in quality of life between participants with and without PPSP | 3 months
  PHQ-8 Score; GAD-7 Score; EQ-5D-5L score at day 97
To investigate the difficulty in reducing opioid use in participants with PPOU | 3 months
  Yes/no question on questionnaire at day 97

OTHER OUTCOMES:
To explore patient experience of; Preparation for day case surgery and pre-operative expectations Acute recovery (first postoperative week) Longer-term recovery and post-operative pain (after 3 months) Opioids: intake, type, duration and experience. | 4-5 months
  Semi-structured questionnaires after day 97, regarding the topics listed above

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rockett, MBBS, PhD, Study Director — University Hospitals Plymouth NHS Trust
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided